CLINICAL TRIAL: NCT05651581
Title: Efficacy and Acceptability of a Monkeypox Curriculum for Disproportionately Impacted Communities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Social Protocol
Record Dates: First submitted 2022-11-26; First posted 2022-12-15 (Actual); Last update posted 2023-10-04 (Actual); Status verified 2023-10

CONDITIONS: Monkey Pox
MeSH Terms: conditions — Mpox, Monkeypox

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Online module — online module including around 5 videos and several infographics covering the topics of symptoms transmission, prevention, vaccination, and treatment of the monkeypox virus.

SUMMARY:
The study team will create an online module via the REDCap platform. The module will include around 5 videos and several infographics covering the topics of symptoms, transmission, prevention, vaccination, and treatment of the monkeypox virus. Surveys assessing the primary and secondary study endpoints will be given to participants before and after the module. The purpose of the study is to assess the efficacy and acceptability of an educational presentation on monkeypox in a cohort of individuals recruited from Rainbow Health and to secondarily assess participant risk perception, intention to vaccinate, and confidence in public health initiatives.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who are 18 years and older
* Individuals able to read and write in English

Exclusion Criteria:

* Unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2023-05-24 (Actual); Primary Completion 2023-08-24 (Actual); Study Completion 2023-08-24 (Actual)

PRIMARY OUTCOMES:
Efficacy of intervention | baseline
  Efficacy of intervention will be measured by changes in knowledge using a survey
Efficacy of intervention | immediately after intervention
  Efficacy of intervention will be measured by changes in knowledge using a survey
Acceptability | immediately after intervention
  Acceptability will be measured by a validated questionnaire based on the Theoretical Framework of Acceptability.

SECONDARY OUTCOMES:
risk perception | baseline
  questionnaire
risk perception | immediately after intervention
  questionnaire
intention to vaccinate | baseline
  questionnaire
intention to vaccinate | immediately after intervention
  questionnaire
confidence in public health initiatives | baseline
  questionnaire
confidence in public health initiatives | immediately after intervention
  questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Mansh, MD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No